CLINICAL TRIAL: NCT00230100
Title: Recovery Group for Women With Substance Use Disorders - Stage I
Brief Title: The Women's Recovery Group Study: Stage I Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Shelly F. Greenfield, Chief Academic Officer, Director, Clinical Research and Education, ADATP, Professor of Psychiatry, McLean Hospital, Harvard Medical School., Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-15434-1; R01DA015434 (NIH)
Record Dates: First submitted 2005-09-29; First posted 2005-09-30 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Alcohol-Related Disorders; Substance-Related Disorders
Keywords: Gender differences; Women; Substance use disorders; Alcohol use disorders; Treatment outcomes; Group therapy
MeSH Terms: conditions — Alcohol-Related Disorders; Substance-Related Disorders; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Women's Recovery Group (Experimental): The Women's Recovery Group (WRG) is a manual-based group therapy for women heterogeneous with respect to their substance use disorder, co-occurring psychiatric disorders, trauma history, age, and stage of life. The WRG is a 12-session, structured relapse-prevention group therapy that utilizes a cognitive behavioral approach and includes gender-specific content and single-gender group composition. Individual session content was derived from research on gender-specific substance abuse antecedents, consequences, and treatment outcomes. The overall goals of the treatment are to (1) promote abstinence from all substances including alcohol; (2) improve understanding of specific aspects of SUDs, recovery, and relapse that are relevant to women, and (3) help participants with skills and strategies useful in preventing relapse and promoting recovery.
  Interventions: Behavioral: The Women's Recovery Group
- mixed-gender Group Drug Counseling (Active Comparator): Group Drug Counseling (GDC) is a standard 12-week, 90-minute mixed-gender group therapy. The overall goals of GDC are to 1) help patients to achieve abstinence from all substances of abuse; 2) educate patients regarding recovery from substance use disorders; 3) increase patients' self-awareness of the problems that their substance use disorder has caused; 4) encourage patients to give mutual support; and 5) help patients learn new ways to cope with problems in order to prevent relapse. The GDC was chosen as the comparison group to approximate group drug counseling that is consistent with treatment as usual within the community.
  Interventions: Behavioral: mixed-gender Group Drug Counseling

INTERVENTIONS:
Behavioral: The Women's Recovery Group — The Women's Recovery Group (WRG) is a manual-based group therapy for women heterogeneous with respect to their substance use disorder, co-occurring psychiatric disorders, trauma history, age, and stage of life. The WRG is a 12-session, structured relapse-prevention group therapy that utilizes a cognitive behavioral approach and includes gender-specific content and single-gender group composition. Individual session content was derived from research on gender-specific substance abuse antecedents, consequences, and treatment outcomes. The overall goals of the treatment are to (1) promote abstinence from all substances including alcohol; (2) improve understanding of specific aspects of SUDs, recovery, and relapse that are relevant to women, and (3) help participants with skills and strategies useful in preventing relapse and promoting recovery.
  Other Names: WRG
  Arms: Women's Recovery Group
Behavioral: mixed-gender Group Drug Counseling — Group Drug Counseling (GDC) is a standard 12-week, 90-minute mixed-gender group therapy. The overall goals of GDC are to 1) help patients to achieve abstinence from all substances of abuse; 2) educate patients regarding recovery from substance use disorders; 3) increase patients' self-awareness of the problems that their substance use disorder has caused; 4) encourage patients to give mutual support; and 5) help patients learn new ways to cope with problems in order to prevent relapse. The GDC was chosen as the comparison group to approximate group drug counseling that is consistent with treatment as usual within the community.
  Other Names: GDC
  Arms: mixed-gender Group Drug Counseling

SUMMARY:
The purpose of this study was to develop a gender-specific 12-session, manual-based relapse prevention group for women with substance use disorders (SUDs).

DETAILED DESCRIPTION:
This Phase I trial compares single-gender Women's Recovery Group (WRG) and an effective control condition, mixed-gender Group Drug Counseling (GDC). WRG is a new 12-session women-focused, manual-based relapse-prevention group therapy that uses a cognitive-behavioral approach. It is a 90-minute structured relapse prevention weekly group therapy with both women-focused content as well as an all-women group composition. The control condition, Group Drug Counseling (GDC), consists of 12 weekly 90-minute structured sessions and is conducted in a mixed-gender group composition and has no women-focused content. The GDC was chosen as the comparison group to approximate group drug counseling that is consistent with treatment as usual within the community. Both groups stress abstinence. Women are randomly assigned to one of the two conditions and the groups are conducted in a rolling group, semi-open format.

The treatment manual for a Women's Recovery Group (WRG) focused on the themes that are relevant to women with SUDs. There was an emphasis on educating patients about treatment and relapse prevention in a context that is relevant to women. The manual combined therapist information and instructions with patient worksheets, handouts and skills practices. The treatment intervention was conducted twice in a pre-pilot study led by study investigators. The investigators then conducted a pilot study in which outcomes among subjects receiving the treatment intervention were compared with outcomes of subjects who received the standard mixed-gender Group Drug Counseling (GDC), chosen to approximate treatment in the community.

The study hypothesis was that the single-gender group composition and women-focused group content would result in better treatment outcomes, including decrease number of days of substance use compared with baseline during follow-up, reduced substance use, and lengthened time to relapse, compared with the mixed-gender control.

ELIGIBILITY:
Inclusion criteria:

Participants were included in the study if they:

* were diagnosed with at least one substance dependence other than nicotine dependence based on the Structured Clinical Interview for DSM-IV at the time of enrollment
* used substances within 60 days of baseline assessment
* were 18 years of age or older
* expressed intention to remain within the geographic area to return for follow-up assessments
* signed permission for the research team to communicate with any other mental health professional from whom they were receiving care

Patients were excluded if they:

* had certain co-occurring diagnoses (i.e., bipolar, post-traumatic stress, or psychotic disorders) at the time of enrollment
* were mandated to treatment
* were in residential treatment restricting substance use during the group treatment phase
* participated in concurrent substance abuse treatment group (not including self-help) during the 12-week group treatment phase
* showed clinical indication for medical detoxification (these patients were eligible to enter the study after detoxification)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-03; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelly F Greenfield, M.D., M.P.H., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Greenfield SF, Trucco EM, McHugh RK, Lincoln M, Gallop RJ. The Women's Recovery Group Study: a Stage I trial of women-focused group therapy for substance use disorders versus mixed-gender group drug counseling. Drug Alcohol Depend. 2007 Sep 6;90(1):39-47. doi: 10.1016/j.drugalcdep.2007.02.009. Epub 2007 Apr 18. PMID 17446014
- [Result] Greenfield SF, Potter JS, Lincoln MF, Popuch RE, Kuper L, Gallop RJ. High psychiatric symptom severity is a moderator of substance abuse treatment outcomes among women in single vs. mixed gender group treatment. Am J Drug Alcohol Abuse. 2008;34(5):594-602. doi: 10.1080/00952990802304980. PMID 18821452
- [Result] McHugh RK, Greenfield SF. Psychiatric Symptom Improvement in Women Following Group Substance Abuse Treatment: Results from the Women's Recovery Group Study. J Cogn Psychother. 2010 Apr 1;24(1):26-36. doi: 10.1891/0889-8391.24.1.26. PMID 20625473
- [Result] Cummings AM, Gallop RJ, Greenfield SF. Self-efficacy and substance use outcomes for women in single gender versus mixed-gender group treatment. J Groups Addict Recover. 2010;5(1):4-16. doi: 10.1080/15560350903543915. PMID 21753920
- [Result] Kuper LE, Gallop R, Greenfield SF. Changes in coping moderate substance abuse outcomes differentially across behavioral treatment modality. Am J Addict. 2010 Nov-Dec;19(6):543-9. doi: 10.1111/j.1521-0391.2010.00074.x. Epub 2010 Sep 23. PMID 20958851
- [Result] Greenfield SF, Cummings AM, Kuper LE, Wigderson SB, Koro-Ljungberg M. A qualitative analysis of women's experiences in single-gender versus mixed-gender substance abuse group therapy. Subst Use Misuse. 2013 Jun;48(9):750-60. doi: 10.3109/10826084.2013.787100. Epub 2013 Apr 22. PMID 23607675
- [Result] Greenfield SF, Kuper LE, Cummings AM, Robbins MS, Gallop RJ. Group Process in the single-gender Women's Recovery Group compared with mixed-gender Group Drug Counseling. J Groups Addict Recover. 2013;8(4):10.1080/1556035X.2013.836867. doi: 10.1080/1556035X.2013.836867. PMID 24294145

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with current substance dependence were recruited from McLean Hospital programs, advertisements, flyers, and clinician referrals. Advertisements were for investigational group therapy for substance abuse but did not specify the Women's Recovery Group in order to minimize selection bias for women only interested in women's treatment.
Pre-assignment Details: Groups were conducted in an semi-open format where enrollment continued until a maximum of 6-8 subjects were entered per group and then enrollment was closed until the end of the sequence.
Period: Overall Study
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Started | 29 | 17
Completed | 29 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling | Total
Number analyzed (Participants) | 29 | 17 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (10.73) | 49.7 (12.5) | 46.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 7 | 36
  Male | 0 | 10 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 29 | 16 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 17 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Days of Any Substance Use for Women
Description: This represents the change from baseline in the mean number of days per month of any substance use (i.e. drug and/or alcohol). Days of substance use was assessed using the Timeline Follow-Back at baseline (assessing for the 60 days prior to the baseline interview) and then monthly for months 1-6 (months 1-3 were in-treatment assessments and months 4-6 were post-treatment follow-up assessments), and month 9 (also a post-treatment follow-up assessment). We implemented a general mixed model analysis of variance (MMANOVA), which models the means per group over the respective time period and the covariance between the repeated measures over the assessments. Both the in-treatment and post-treatment time frames were compared to baseline substance use data.
Time Frame: In-treatment phase (month 1-3), Post-treatment phase (month 4-6, 9)
Population: Only women were included in this analysis.
Measure: Mean (Standard Error); unit: Days of any substance use per month
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 29 | 7
Days of any substance use per month
  In-treatment Phase (months 1-3) | -3.93 (1.35) | -1.74 (3.07)
  Post-treatment Phase (month 4-6, 9) | -4.45 (1.32) | 0.60 (3.02)
Statistical Analysis 1: Comparison: Women's Recovery Group vs Mixed-gender Group Drug Counseling; Implemented a general mixed model analysis of variance (MMANOVA), which models the means per group over the respective time period and the covariance between the repeated measures over the assessments. The MMANOVA approach estimates a separate mean for each phase of treatment per group. The MMANOVA is called a "mixed" model because it includes both fixed (e.g., treatment, gender) and random (subject-specific) terms. MMANOVA allows for randomly missing observations (not included in analysis); Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

2. Primary Outcome: Change in Mean Number of Drinking Days for Women
Description: This represents the change from baseline in the mean number of drinking days for women. Number drinking days was assessed using the Timeline Follow-Back at baseline (assessing for the 60 days prior to the baseline interview) and then monthly for months 1-6 (months 1-3 were in-treatment assessments and months 4-6 were post-treatment follow-up assessments), and month 9 (also a post-treatment follow-up assessment). We implemented a general mixed model analysis of variance (MMANOVA), which models the means per group over the respective time period and the covariance between the repeated measures over the assessments. Both the in-treatment and post-treatment time frames were compared to baseline substance use data.
Time Frame: In-treatment phase (month 1-3), Post-treatment phase (month 4-6, 9)
Population: Only women were included in this analysis.
Measure: Mean (Standard Error); unit: Drinking days
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 29 | 7
Drinking days
  In-treatment Phase (months 1-3) | -1.95 (0.98) | -0.23 (2.23)
  Post-treatment Phase (month 4-6, 9) | -2.40 (0.95) | 1.72 (2.17)
Statistical Analysis 1: Comparison: Women's Recovery Group vs Mixed-gender Group Drug Counseling; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

3. Secondary Outcome: Change in Mean Number of Drinks Per Drinking Day for Women
Description: This represents the change from baseline in the mean number of drinks per drinking day for women. The number of drinks per drinking day was measured using the Timeline Follow-Back at baseline (assessing for the 60 days prior to the baseline interview) and then monthly for months 1-6 (months 1-3 were in-treatment assessments and months 4-6 were post-treatment follow-up assessments), and month 9 (also a post-treatment follow-up assessment). We implemented a general mixed model analysis of variance (MMANOVA), which models the means per group over the respective time period and the covariance between the repeated measures over the assessments. Both the in-treatment and post-treatment time frames were compared to baseline substance use data.
Time Frame: In-treatment phase (month 1-3), Post-treatment phase (month 4-6, 9)
Population: Only women were included in this analysis.
Measure: Mean (Standard Error); unit: Drinks per drinking day
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 29 | 7
Drinks per drinking day
  In-treatment Phase (months 1-3) | -0.62 (0.72) | 0.36 (1.64)
  Post-treatment Phase (month 4-6, 9) | -1.19 (0.71) | 1.66 (1.62)
Statistical Analysis 1: Comparison: Women's Recovery Group vs Mixed-gender Group Drug Counseling; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

4. Secondary Outcome: Change in Mean Addiction Severity Index Alcohol Composite Score for Women
Description: This represents the change from baseline in mean composite scores of the Addiction Severity Index (ASI) alcohol section. The ASI was administered at baseline (assessing for the 60 days prior to the baseline interview) and then monthly for months 1-6 (months 1-3 were in-treatment assessments and months 4-6 were post-treatment follow-up assessments), and month 9 (also a post-treatment follow-up assessment). We implemented a general mixed model analysis of variance (MMANOVA), which models the means per group over the respective time period and the covariance between the repeated measures over the assessments. Both the in-treatment and post-treatment time frames were compared to baseline substance use data.
  The ASI is a widely employed multidimensional assessment of substance-related problems. Scores range from 0-1 where higher scores reflect higher addiction severity.
Time Frame: In-treatment phase (month 1-3), Post-treatment phase (month 4-6, 9)
Population: Only women were included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 29 | 7
units on a scale
  In-treatment Phase (months 1-3) | -0.14 (0.04) | -0.14 (0.10)
  Post-treatment Phase (month 4-6, 9) | -0.23 (0.04) | -0.03 (0.10)
Statistical Analysis 1: Comparison: Women's Recovery Group vs Mixed-gender Group Drug Counseling; It was hypothesized that the single-gender group composition and women-focused group content (WRG) would result in better substance abuse treatment outcomes (lower ASI alcohol composite scores) than standard mixed-gender group treatment (GDC); Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

5. Post Hoc Outcome: Client Satisfaction for Women
Description: Participant satisfaction with the groups was assessed using the Client Satisfaction Questionnaire (CSQ-8) plus four additional questions about the helpfulness of the therapist, group content, and group composition. Questions were answered on a 4-point scale where 1 reflected negative feelings and 4 reflected positive feelings. Participants' scores are calculated by adding up the numbers assigned to their chosen answers. Therefore, scores can range between 12 and 48, with higher scores reflecting greater satisfaction.
  The CSQ was administered at week 3, 6, 9, and 12 while participants were in treatment. Scores represent calculated averages of the group averages for week 3, week 6, week 9, and week 12.
Time Frame: In treatment phase (week 1-12)
Population: Only women were included in this analysis.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 29 | 7
units on a scale | 44.49 [43.13 to 45.46] | 40.44 [38.00 to 43.75]
Statistical Analysis 1: Comparison: Women's Recovery Group vs Mixed-gender Group Drug Counseling; Test type: Superiority or Other; p < 0.009, Mixed Models Analysis

6. Other Pre Specified Outcome: Baseline Substance Use Data for Women
Description: The data reflect baseline characteristics of women participants with respect to (1) days of any substance use (i.e. drugs or alcohol), and (2) the number of drinking days, in the 60 days prior to baseline intake.This data was collected using the Timeline Follow-Back.
Time Frame: Baseline
Population: Only women were included in this analysis.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 29 | 7
Days
  Days of any substance use | 13.17 (1.87) | 11.09 (2.11)
  Number of drinking days | 10.38 (1.42) | 10.23 (1.80)

7. Other Pre Specified Outcome: Baseline Drinks Per Drinking Day for Women
Description: The data reflect baseline characteristics of the women participants with respect to the number of drinks per drinking day in the 60 days prior to baseline intake. This was measured using the Timeline Follow-Back.
Time Frame: Baseline
Population: Only women were included in this analysis.
Measure: Mean (Standard Error); unit: Drinks per drinking day
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 29 | 7
Drinks per drinking day | 6.56 (0.93) | 6.14 (1.18)

8. Other Pre Specified Outcome: Baseline Addiction Severity Index Alcohol Composite Score for Women
Description: The data reflect baseline characteristics of the participants with respect to ASI alcohol composite score. Scores range between 0 and 1. Higher scores reflect higher addiction severity. The ASI is a multidimensional assessment of substance-related problems which yields composite scores for alcohol use, drug use, psychiatric status, medical status, legal status, family/social relationships, and employment status.
Time Frame: Baseline
Population: Only women were included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Number analyzed (Participants) | 29 | 7
units on a scale | 0.45 (0.05) | 0.44 (0.11)

ADVERSE EVENTS:
Time Frame: Weekly from weeks 1-12 (in treatment)
Description: Both women and men are included.
Groups:
- Women's Recovery Group: The WRG is a manual-based group therapy for women heterogeneous with respect to their substance dependence, co-occurring psychiatric disorders, trauma history, and age and stage of life. The WRG is a 12-session, structured relapse-prevention group therapy that utilizes a cognitive behavioral approach and includes gender-specific content and single-gender group composition. Individual session content was derived from research on gender-specific substance abuse antecedents, consequences, and treatment outcomes. The overall goals of the treatment are to (1) promote abstinence from all substances including alcohol; (b) improve understanding of specific aspects of SUDs, recovery, and relapse that are relevant to women, and (c) help participants with skills and strategies useful in preventing relapse and promote recovery.
- Mixed-gender Group Drug Counseling: The GDC is a standard 12-week, 90-minute mixed-gender group therapy. The overall goals of GDC are to 1) help patients to achieve abstinence from all substances of abuse; 2) educate patients regarding recovery from substance dependence; 3) increase patients' self-awareness of the problems that substance dependence has caused; 4) encourage patients to give mutual support; and 5) help patients learn new ways to cope with problems in order to prevent relapse.
Arm/Group | Women's Recovery Group | Mixed-gender Group Drug Counseling
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/17
Other Adverse Events (participants affected / at risk) | 0/29 | 0/17

LIMITATIONS AND CAVEATS:
* small sample
* small proportion had drug dependence; majority had alcohol dependence (questionable generalizability)
* sample was almost all white and well-educated (questionable generalizability)
* therapists not blind to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes